CLINICAL TRIAL: NCT00247130
Title: A Prospective, Randomized Trial Comparing the Effect of Intravenous Omeprazole to That of Intravenous Ranitidine on the Maintenance of Hemostasis After Successful Endoscopic Treatment of Bleeding Peptic Ulcer
Brief Title: Comparison of Intravenous Omeprazole to Ranitidine on Recurrent Bleeding After Endoscopic Treatment of Bleeding Ulcer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Superiority of iv omeprazole to ranitidine has already been proven by others.
Sponsor: Keio University (Other)
Responsible Party: Principal Investigator, Hidekazu Suzuki, M.D., Ph.D., Associate Professor, Keio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KEIO-UGI-001
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Peptic Ulcers
Keywords: Omeprazole; Ranitidine; Endoscopic treatment; Hemostasis; Peptic ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — Omeprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator): Omeprazole (20 mg), intravenous, 2x /day
  Interventions: Drug: Omeprazole
- Ranitidine (Active Comparator): Ranitidine (100 mg), intravenous drip infusion, 2x /day.
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Omeprazole
  Other Names: omeprazon
  Arms: Omeprazole
Drug: Ranitidine
  Other Names: Zantac
  Arms: Ranitidine

SUMMARY:
The present study will compare the hemostasis-maintaining effects of intravenous omeprazole and ranitidine in patients with upper gastrointestinal hemorrhage that have undergone endoscopic hemostasis, to establish which anti-secretory medication prior to the start of oral alimentation is effective in preventing re-hemorrhage after hemostasis.

DETAILED DESCRIPTION:
Gastrointestinal hemorrhage is a relatively common condition, with the source of the bleeding being most commonly from the upper gastrointestinal tract, especially from gastric and duodenal ulcers. It often requires emergency treatment. First, the site of bleeding is determined. If an exposed blood vessel is found in the hemorrhagic lesion, or in the case of oozing or projectile hemorrhage, endoscopic hemostasis is performed on the lesion. After hemostasis is achieved, prevention of re-bleeding is important; usually, an antacid or similar medication is administered and the course is monitored under fasting conditions.Suppression of gastric acid secretion is necessary to raise gastric pH levels and maintain normal blood coagulation, and to promote healing of hemorrhagic lesions. In Japan, intravenous preparations of H2 receptor antagonists and proton pump inhibitors have been commonly used.In foreign countries, drug therapy for patients with upper gastrointestinal hemorrhage emphasizes the maintenance of normal blood coagulation. High doses of these drugs have been established to constantly maintain a pH of 7 in the stomach (Daneshmend TK, et al., BMJ 1992, 304:143-147; Labentz J, et al., Gut 1997, 40:36-41; Hasselgren G, et al., Scand J Gastroenterol 1997, 32:328-333; Schaffalitzky de Muckadell OB, et al., Scand J Gastroenterol 1997, 32:320-327; Sung JJY, et al., Ann Intern Med 2003, 139:237-243). In a clinical study, proton pump inhibitors were superior to H2 receptor antagonists in terms of clinical efficacy (Labentz J, et al., Gut 1997, 40:36-41). In Japan, emphasis is placed on promoting healing of lesions since endoscopic hemostasis is a fairly common practice; doses have been established at levels similar to therapeutic doses for peptic ulcers. It cannot be said, however, that superiority of intravenous proton pump inhibitors over H2 receptor antagonists has been established at such doses. This can possibly be attributed to fact that in previous studies the study populations were not homogenous in terms of severity; for example, patients requiring endoscopic hemostasis and those that did not were both included.Against this background, this study will compare the hemostasis-maintaining effects of intravenous omeprazole and ranitidine in patients with upper gastrointestinal hemorrhage that have undergone endoscopic hemostasis, to establish which anti-secretory medication prior to the start of oral alimentation is effective in preventing re-hemorrhage after hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with identified gastric or duodenal ulcer
* Patients with hemorrhagic exposed vessel at the ulcer lesion, oozing or projectile hemorrhage (predominantly arterial) from the ulcer, and where endoscopic hemostasis has been performed.
* Over 20 years of age of either sex.
* The subject or his or her proxy consenter has provided written informed consent.

Exclusion Criteria:

* Serious hepatopathy, nephropathy, or heart disease.
* Complicating malignant tumor.
* Hemorrhage from malignant tumor.
* The patient is on, or in need of, treatment with a drug considered to interact with the test drug.
* History of allergy to the test drug.
* History of anaphylactic shock.
* Pregnant, possibly pregnant, or lactating.
* patient who is unable to fully understand the explanation about the study.
* patient who is judged by the investigator to be otherwise inappropriate for inclusion.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
No evidence of hemorrhage or vessel exposure on a second endoscopy | 4 weeks after the bleeding

SECONDARY OUTCOMES:
Plasma ghrelin levels | 4 weeks after the bleeding
Serum gastrin levels | 4 weeks after the bleeding
No evidence of hemorrhage or vessel exposure on a third endoscopy | 12 weeks after the bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, M.D., Ph.D., Study Chair — Division of Gastroenterology, Department of Internal Medicine, Keio University School of Medicine; Hidekazu Suzuki, M.D., Ph.D., Principal Investigator — Upper GI Research Center, Keio University School of Medicine
Locations (1):
- Department of Internal Medicine, Keio University School of Medicine, Tokyo, Tokyo, Japan